CLINICAL TRIAL: NCT06629987
Title: Determining the Most Efficient Screening Cut Off Levels for Phenylketonuria (PKU) by Assessing Two Years of Screening with Tandem Mass Spectrometry (MS) : a French National Cohort Study
Brief Title: Determining the Most Efficient Screening Cut Off Levels for Phenylketonuria (PKU)
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University Hospital, Lille (Other); Hospices Civils de Lyon (Other); University Hospital, Strasbourg, France (Other); CHU de Reims (Other); Centre Hospitalier Universitaire, Amiens (Other); Centre Hospitalier Universitaire Dijon (Other); Nantes University Hospital (Other); University Hospital, Tours (Other); Clinical Research Center of Reunion island (Unknown); University Hospital, Caen (Other); Rennes University Hospital (Other); University Hospital, Bordeaux (Other); University Hospital, Toulouse (Other); University Hospital, Montpellier (Other)
Responsible Party: Principal Investigator, HESS Valentin, MD, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2022PI186
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: PKU
Keywords: screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
studying the screening of PKU in france with the new tandemMS

DETAILED DESCRIPTION:
Nationwide cohort study of the new pku screening for patient beetwen 180 and 360 µmol/L.

ELIGIBILITY:
Inclusion Criteria:

* having screening in france

Exclusion Criteria:

* refusing neonatal screening

Min Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all french population born who had a screening
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
developping an PKU: id phenylanine over 360µmol/L | 1 year
  based on level of phenylalanine during the year of follow up

SECONDARY OUTCOMES:
screening value | 2 years
  determining the bets screening value

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU NANCY hopital enfant, Nancy, France